CLINICAL TRIAL: NCT01420744
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel-group, Adaptive Group-sequential Phase II Study, to Determine the Efficacy and Safety of BT086 as an Adjunctive Treatment in Severe Community Acquired Pneumonia (sCAP)
Brief Title: Safety and Efficacy Study of BT086 to Evaluate Adjunctive Therapy in sCAP
Acronym: CIGMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIGMA Study 982
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Community Acquired Pneumonia
Keywords: Endotracheal ventilation; Bacterial pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BT086 infusion (Experimental)
  Interventions: Drug: BT086
- 1% Human Albumin infusion (Placebo Comparator)
  Interventions: Drug: 1% Human Albumin infusion

INTERVENTIONS:
Drug: BT086 — BT086 will be administered per intravenous infusion (IV). The dose to be administered is 3.65 mL /kg bw/day and is calculated by the mean Immunoglobulin M (IgM) content of BT086 which is 23%.
  Infusion rate:
  Starting rate is 0.1 mL/min. Maximum infusion rate is 0.5 mL/min (target infusion rate) Treatment will be administered over a 5-day period.
  Arms: BT086 infusion
Drug: 1% Human Albumin infusion — 1% Albumin will be administered per intravenous infusion (IV). The dose to be administered is 3.65 mL /kg bw/day.
  Infusion rate:Starting rate is 0.1 mL/min. Maximum infusion rate is 0.5 mL/min (target infusion rate). Rate is to be raised in steps of 0.1 mL every 10 min until the target infusion rate is reached.
  Treatment will be administered over a 5-day period.
  Starting rate is 0.1 mL/min. Maximum infusion rate is 0.5 mL/min (target infusion rate)
  Arms: 1% Human Albumin infusion

SUMMARY:
The purpose of this study is to determine whether the adjunctive therapy to standard antibiotic treatment of BT086 is safe and effective of decreasing the days patients require endotracheal ventilation due to Severe Community-Acquired Pneumonia (sCAP).

DETAILED DESCRIPTION:
Severe Community-Acquired Pneumonia (sCAP) is usually defined clinically as pneumonia acquired from outside the hospital (CAP) that requires intensive medical care. Mortality of (s)CAP patients admitted to ICU range from 35-58% depending on time and admission of the patient and has not much improved in the last years.

BT086 contains a sufficient number of antibodies against the most frequent pathogens as well as antibodies against lipopolysaccharides and lipid A. Therefore, it can be assumed that administration of BT086 early in the clinical course of a severe infection such as sCAP may provide an effective adjunctive treatment to standard antibiotic therapy for sCAP patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent:

  * given by the patient or
  * a legal/authorised representative of the patient or
  * a waiver for written informed consent due to emergency situation, in compliance with all local legal requirements.
* Male or female patients aged 18 years or older
* Patient receiving adequate antibiotic treatment for pneumonia
* Prior to endotracheal ventilation and therapy, the patient must have at least one of the following two signs of inflammation:

  * Fever/Hypothermia Fever defined as an oral, tympanic, oesophageal or vesical temperature of >38°C, tympanic temperature of >38°C or rectal temperature of >38.5°C, or hypothermia (rectal temperature <35.5°C) (measurement with temperature probe or device) or
  * White blood cell (WBC) count >10,000/mm³ or WBC <4,500/mm³
* Patient must have at least one of the following signs and symptoms of pneumonia:

  * New or increased cough
  * Production of purulent sputum or change in sputum characteristics
  * Dyspnoea or tachypnoea (respiratory rate >20 breaths/minute)
  * Pleuritic chest pain
  * Auscultatory findings on pulmonary examination of rales and/or crackles and/or evidence of pulmonary consolidation (e.g. dullness on percussion, bronchial breath sounds, or egophony)
* Radiological (or other imaging technique) evidence of (an) infiltrate(s) consistent with bacterial pneumonia
* Pneumonia has been acquired outside the hospital. In hospital-admitted patients, pneumonia has been diagnosed a maximum of 72 hours after admission. Patients from nursing homes or similar institutions are eligible.
* Major sCAP criterion: need for endotracheal ventilation
* Treatment of patient with BT086 must start within 12 hours but not earlier than 1 hour after start of endotracheal ventilation

Exclusion Criteria:

* For incapacitated patients: any indication that the patient's presumed will would be against inclusion in the trial
* Patients with suspected hospital-acquired pneumonia
* Severe lung diseases interfering with sCAP therapy e.g. patients with cystic fibrosis,
* Patients receiving Xigris® (drotrecogin alfa, activated Protein C) or medications not approved for sCAP (e.g. Dornase alpha) are excluded from inclusion in the study
* Patients on dialysis
* Presence of other severe diseases impairing life expectancy (e.g. patients are not expected to survive 28 days given their pre-existing uncorrectable medical condition).
* Patients unable to be treated due to obesity
* Selective, absolute IgA deficiency with known antibodies to IgA
* Patients with neutrophil count <1,000/mm³ or platelet count <50,000/mm³
* Pregnant or lactating women. A pregnancy test will be performed in all women aged <65 years and the result must be available at study inclusion.
* Known relevant intolerance to immunoglobulins, vaccines or other substances of human origin
* Participation in another interventional clinical trial within 30 days before entering the study or during the study, and/or previous participation in this study (participation in non-interventional trials is allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-08; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Ventilator Free Days (VFDs) | 28 days
  VFDs are defined as the number of days between successful weaning from endotracheal ventilation and day 28 after study enrolment.

SECONDARY OUTCOMES:
28-day all cause mortality | 28 days (672 hours from randomization)
  All patients will be classified as either "alive at Study Day 28" or, if dead, "dead at Study Day 28", regardless of cause of death.
28-day pneumonia-cause mortality | 28 days (672 hours from randomization)
  All patients will be classified as either "alive at Study Day 28" or, if dead, "dead at Study Day 28, with pneumonia as cause of death".
Time (days) to discharge from ICU | 28 days
  The date and time of admission to and discharge from the ICU will be recorded in the Case Report Form (CRF). The time to discharge from the ICU will be calculated as the number of days spent in the ICU.
Time (days) to discharge from hospital | 28 days
  The date and time of admission to and discharge from the hospital will be recorded in the CRF. The time to discharge from the hospital will be calculated as the number of days spent in the hospital.
SOFA: Score Sequential Organ Failure Assessment | 28 days
  Each organ system (cardiovascular, haematology, hepatic, renal, respiratory) will be scored using the SOFA methodology.For analysis, a patient will receive a score on each day (Study Days 1-7, Day 14, Day 21, and Day 28). Mean changes in organ function scores over time and percentages of patients whose organ function has resolved will be compared between treatment groups.
Vasopressor-free days | 28 days
  Vasopressor-free days will be calculated in a similar manner to VFDs, as described above. Vasopressors include dobutamine, epinephrine, dopamine, and norepinephrine.
  A day is considered as a vasopressor-free day if a patient does not receive
  * Dobutamine >2.5 µg/kg/min or/and
  * Epinephrine (adrenalin) >=2.5 µg/min or/and
  * Dopamine >=2.5 µg/kg/min or/and
  * Norepinephrine >=0.014 µg/kg/min for 4 hours per day.
Glasgow Coma Score | 28 days
  The Glasgow Coma Scale will be scored using the Glasgow Coma Score methodology. The patient will be assessed by calculating the score on each study day (Day -1 through to Day 28).

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Welte, MD, Principal Investigator — Hannover Medical School
Locations (36):
- 401, Brussels, Belgium
- Germany (17):
  - 108, Berlin
  - 114, Chemnitz
  - 118, Cologne
  - 119, Cologne
  - 110, Dresden
  - 111, Erfurt
  - 116, Frankfurt
  - 117, Greifswald
  - 103, Halle
  - 115, Hamburg
  - 101, Hanover
  - 107, Homburg/Saar
  - 109, Lübeck
  - 106, Marburg
  - 120, Stuttgart
  - 105, Tübingen
  - 113, Wuppertal
- Spain (12):
  - 213, Badalona
  - 201, Barcelona
  - 206, Barcelona
  - 204, Girona
  - 207, Madrid
  - 208, Mataró
  - 210, Palma de Mallorca
  - 212, Sabadell
  - 209, Santiago de Compostela
  - 205, Tarragona
  - 211, Terrassa
  - 203, Valencia
- United Kingdom (6):
  - 303, Cardiff
  - 304, Kings Lynn, Norfolk
  - 301, London
  - 306, London
  - 302, Poole, Dorset
  - 305, Reading, Berkshire

REFERENCES:
- [Derived] Jahn K, Handtke S, Palankar R, Weissmuller S, Nouailles G, Kohler TP, Wesche J, Rohde M, Heinz C, Aschenbrenner AF, Wolff M, Schuttrumpf J, Witzenrath M, Hammerschmidt S, Greinacher A. Pneumolysin induces platelet destruction, not platelet activation, which can be prevented by immunoglobulin preparations in vitro. Blood Adv. 2020 Dec 22;4(24):6315-6326. doi: 10.1182/bloodadvances.2020002372. PMID 33351126
- [Derived] Welte T, Dellinger RP, Ebelt H, Ferrer M, Opal SM, Singer M, Vincent JL, Werdan K, Martin-Loeches I, Almirall J, Artigas A, Ignacio Ayestaran J, Nuding S, Ferrer R, Sirgo Rodriguez G, Shankar-Hari M, Alvarez-Lerma F, Riessen R, Sirvent JM, Kluge S, Zacharowski K, Bonastre Mora J, Lapp H, Wobker G, Achtzehn U, Brealey D, Kempa A, Sanchez Garcia M, Brederlau J, Kochanek M, Reschreiter HP, Wise MP, Belohradsky BH, Bobenhausen I, Dalken B, Dubovy P, Langohr P, Mayer M, Schuttrumpf J, Wartenberg-Demand A, Wippermann U, Wolf D, Torres A. Efficacy and safety of trimodulin, a novel polyclonal antibody preparation, in patients with severe community-acquired pneumonia: a randomized, placebo-controlled, double-blind, multicenter, phase II trial (CIGMA study). Intensive Care Med. 2018 Apr;44(4):438-448. doi: 10.1007/s00134-018-5143-7. Epub 2018 Apr 9. PMID 29632995